CLINICAL TRIAL: NCT07097363
Title: A Pilot Study of Epcoritamab With Dose Adjusted Etoposide, Cyclophosphamide, Vincristine, Doxorubicin, Prednisone and Rituximab (EPOCH-R) for Upfront Treatment of Aggressive B-Cell Non-Hodgkin Lymphomas
Brief Title: Epcoritamab With Dose Adjusted Etoposide, Cyclophosphamide, Vincristine, Doxorubicin, Prednisone and Rituximab (EPOCH-R) for the Treatment of Aggressive B-Cell Non-Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1125011; NCI-2025-04889 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20955 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2025-07-23; First posted 2025-07-31 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: B-Cell Non-Hodgkin Lymphoma; Burkitt Lymphoma; Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; EBV-Positive Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; High Grade B-Cell Lymphoma With MYC and BCL2 and/or BCL6 Rearrangements; High Grade B-Cell Lymphoma, Not Otherwise Specified; Primary Mediastinal Large B-Cell Lymphoma; T-Cell/Histiocyte-Rich Large B-Cell Lymphoma; Transformed B-Cell Lymphoma, Unclassifiable, With Features Intermediate Between Diffuse Large B-Cell Lymphoma and Classic Hodgkin Lymphoma to Diffuse Large B-Ce
MeSH Terms: conditions — Lymphoma, B-Cell; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — Specimen Handling; Biopsy; Cyclophosphamide; Doxorubicin; Etoposide; Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy; Prednisone; deltacortene; prednylidene; Rituximab; CT-P10

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Epcoritamab and EPOCH-R) (Experimental): Patients receive rituximab IV on day 1, prednisone PO BID on days 1-5, etoposide IV and doxorubicin on days 1-4 and cyclophosphamide IV on day 5 of each cycle. Patients also receive epcoritamab SC on days 8 and 15 of cycle 1, days 1, 8 and 15 of cycles 2-4 and day 1 of cycles 5-6. Cycles repeat every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo MUGA scan or echocardiography during screening and receive fludeoxyglucose and undergo PET scan, CT scan, bone marrow biopsy and aspirate (if needed), and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Doxorubicin; Procedure: Echocardiography Test; Biological: Epcoritamab; Drug: Etoposide; Other: Fludeoxyglucose F-18; Procedure: Multigated Acquisition Scan; Procedure: Positron Emission Tomography; Drug: Prednisone; Biological: Rituximab

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
Procedure: Echocardiography Test — Undergo echocardiography
  Other Names: EC; Echocardiography
Biological: Epcoritamab — Given SC
  Other Names: Anti-CD20/CD3 Bispecific Antibody GEN3013; DuoBody-CD3xCD20; Epcoritamab-bysp; Epkinly; GEN 3013; GEN-3013; GEN3013; Tepkinly
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
Other: Fludeoxyglucose F-18 — Given fludeoxyglucose
  Other Names: 18FDG; FDG; Fludeoxyglucose (18F); fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Procedure: Multigated Acquisition Scan — Undergo MUGA scan
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Biological: Rituximab — Given IV
  Other Names: ABP 798; ABP-798; ABP798; BI 695500; BI-695500; BI695500; Blitzima; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT P10; CT-P10; CTP10; GP 2013; GP-2013; GP2013; IDEC 102; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; IDEC102; Ikgdar; Mabtas; MabThera; Monoclonal Antibody IDEC-C2B8; PF 05280586; PF-05280586; PF05280586; Riabni; Ritemvia; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar GP2013; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; Rituximab-abbs; Rituximab-arrx; Rituximab-blit; Rituximab-pvvr; Rituximab-rite; Rituximab-rixa; Rituximab-rixi; Rixathon; Riximyo; RTXM 83; RTXM-83; RTXM83; Ruxience; Truxima

SUMMARY:
This phase II trial tests the safety, best dose, and effectiveness of epcoritamab when given with etoposide, cyclophosphamide, vincristine, doxorubicin, prednisone and rituximab (EPOCH-R) for the treatment of patients with aggressive B-cell non-Hodgkin lymphoma. Epcoritamab is a bispecific antibody that can bind to two different antigens at the same time. Epcoritamab binds to CD3, a T-cell surface antigen, and CD20 (a tumor-associated antigen that is expressed on B-cells during most stages of B-cell development and is often overexpressed in B-cell cancers) and may interfere with the ability of cancer cells to grow and spread. Etoposide is in a class of medications known as podophyllotoxin derivatives. It blocks a certain enzyme needed for cell division and DNA repair and may kill cancer cells. Cyclophosphamide is in a class of medications called alkylating agents. It works by damaging the cell's DNA and may kill cancer cells. It may also lower the body's immune response. Vincristine is in a class of medications called vinca alkaloids. It works by stopping cancer cells from growing and dividing and may kill them. Doxorubicin is in a class of medications called anthracyclines. Doxorubicin damages the cell's DNA and may kill cancer cells. It also blocks a certain enzyme needed for cell division and DNA repair. Prednisone is in a class of medications called corticosteroids. It is used to reduce inflammation and lower the body's immune response to help lessen the side effects of chemotherapy drugs. Rituximab is a monoclonal antibody. It binds to a protein called CD20, which is found on B cells (a type of white blood cell) and some types of cancer cells. The EPOCH-R is administrated as the standard of care treatment. This may help the immune system kill cancer cells. Giving epcoritamab with EPOCH-R may be safe, tolerable, and effective in treating patients with aggressive B-cell non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive rituximab intravenously (IV) on day 1, prednisone orally (PO) twice daily (BID) on days 1-5, etoposide IV and doxorubicin on days 1-4 and cyclophosphamide IV on day 5 of each cycle. Patients also receive epcoritamab subcutaneously (SC) on days 8 and 15 of cycle 1, days 1, 8 and 15 of cycles 2-4 and day 1 of cycles 5-6. Cycles repeat every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo multigated acquisition (MUGA) scan or echocardiography during screening and receive fludeoxyglucose and undergo positron emission tomography (PET) scan, computed tomography (CT) scan, bone marrow biopsy and aspirate (if needed), and blood sample collection throughout the study.

After completion of study treatment, patients are followed up periodically for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Untreated aggressive large-B cell lymphoma (non-Hodgkin lymphoma) with adverse features that may predict sub-optimal response to R-CHOP and in the opinion of the investigator would be treated with dose adjusted (DA)-EPOCH-R as standard of care. Subjects must be planned to receive full course (6 cycles) chemoimmunotherapy as per clinical standard of care. 1 prior cycle of chemoimmunotherapy may be allowed. Composite lymphomas are not excluded provided that the subject has not received prior systemic therapy for the indolent component and would receive DA-EPOCH-R as the standard of care regimen for the aggressive component. Eligible histologies based on 2016 World Health Organization (WHO) classification include:

  * High grade B-cell lymphoma with MYC and BCL2 and/or BCL6 translocations
  * High grade B-cell lymphoma, not otherwise specified (NOS)
  * Diffuse large b-cell lymphoma (DLBCL) NOS
  * Primary mediastinal B-cell lymphoma
  * T-cell/histiocyte-rich large-B-cell lymphoma
  * Epstein Barr virus (EBV) + DLBCL, NOS
  * Burkitt lymphoma
  * B-cell lymphoma, unclassifiable, with features intermediate between DLBCL and classical Hodgkin lymphoma
* Be willing and able to provide written informed consent for the trial
* Be ≥ 18 years of age on day of signing informed consent
* Have measurable disease, including at least 1 nodal site measuring 1.5 cm or 1 extranodal site measuring 1.0 cm in longest dimension on CT or FDG-PET
* Have a performance status of 0-2 on the Eastern Cooperative Oncology Group (ECOG) performance scale (PS) at time of enrollment
* Left ventricular ejection fraction (LVEF) ≥ 50% on cardiac multiple-gated acquisition (MUGA) scan or cardiac echocardiogram (ECHO)
* Absolute neutrophil count (ANC) ≥ 1,000/μL except in cases of marrow infiltration by lymphoma
* Platelets ≥ 75,000 / mcL except in cases of marrow infiltration by lymphoma or hypersplenism
* Hemoglobin ≥ 8 g/dL except in cases of marrow infiltration by lymphoma without red blood cell (RBC) transfusion within 14 days of first treatment
* Measured or calculated* creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine clearance [CrCl]) ≥ 45 mL/min

  * Creatinine clearance should be calculated per institutional standard
* Serum total bilirubin ≤ 1.5 X upper limit of normal (ULN) (Patients with documented Gilbert disease may be enrolled if total bilirubin ≤ 3.0 x ULN) OR direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver involvement
* International Normalized Ratio (INR) ≤ 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants or prothrombin Time (PT) ≤ 1.5 X ULN unless subject is receiving anticoagulant therapy
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of ≤ 1% per year during the treatment period and for at least 12 months after the last dose of study treatment. Women must refrain from donating eggs during this same period. A woman is considered to be of childbearing potential if she is post-menarcheal, has not reached a postmenopausal state (≤ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). The definition of childbearing potential may be adapted for alignment with local guidelines or requirements. Examples of contraceptive methods with a failure rate of ≤ 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not acceptable methods of contraception
* For women of childbearing potential, a negative serum pregnancy test result during screening period. Women who are considered not to be of childbearing potential are not required to have a pregnancy test
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm, as defined below: With female partners of childbearing potential or pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 6 months after the last treatment. Men must refrain from donating sperm during this same period. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of preventing drug exposure. Male patients considering preservation of fertility should bank sperm before study treatment

Exclusion Criteria:

* Contraindication to any of the individual components of EPOCH-R, including, or history of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies, or known sensitivity or allergy to murine products or if receiving an additional 6 cycles of anthracycline would place patient over the anthracycline lifetime cumulative dose (400 mg/m^2)
* Prior systemic treatment for lymphoma. Prior radiotherapy is allowed provided that this site is not used as a measurable site to assess response
* Transformation from indolent lymphoma is allowed provided that the subject has not received prior systemic therapy for their lymphoma and the aggressive component meets one of the criteria listed in inclusion criterion
* Prior organ transplantation
* Current grade > 1 peripheral neuropathy by clinical examination or demyelinating form of Charcot-Marie-Tooth disease
* Prior systemic therapy for indolent lymphoma
* Prior therapy for large B-cell lymphoma except for patients who require lymphoma symptom control during screening may receive steroids and/or 1 cycle of chemoimmunotherapy in the following manner:

  * Up to 30 mg/day of prednisone or equivalent may be used for lymphoma symptom control during screening, including prior to finalization of staging (not included as part of pre-phase treatment). If glucocorticoid treatment is urgently required at higher doses for lymphoma symptom control prior to the start of study treatment, tumor assessments must be completed prior to initiation of > 30-100 mg/day of prednisone or equivalent. Prednisone > 30-100 mg/day or equivalent may be given for a maximum of 7 days as a pre-phase treatment. If patients exceed the allowed dosing of corticosteroids, patients may still be eligible for the study provided that baseline imaging is performed (or repeated) after completion of the course of higher dose of steroids. Allowed corticosteroid dosing resets from the point of imaging forward and patients who do not exceed the allowed corticosteroid dosing from the point of imaging until initiation of study treatment may enroll. A maximum of 1 cycle of chemoimmunotherapy is allowed if needed for urgent disease stabilization if patient had staging PET/CT and LVEF evaluation prior to chemoimmunotherapy; in this situation patients will receive therapy on study starting with C1D8 epcoritamab provided the next cycle of EPOCH-R chemotherapy will not be delayed by > 7 days
* History of other malignancy that could affect compliance with the protocol or interpretation of results except with permission of the principal investigator. The following are eligible without a specific waiver:

  * Patients with a history of curatively treated basal or squamous cell carcinoma or melanoma of the skin or in situ carcinoma of the cervix at any time prior to the study are eligible.
  * Patients with any malignancy appropriately treated with curative intent and the malignancy has been in remission without treatment for ≥ 2 years prior to enrollment are eligible.
  * Patients with low-grade, early-stage prostate cancer (Gleason score 6 or below, stage 1 or 2) with no requirement for therapy at any time prior to study are eligible
* Evidence of significant, uncontrolled, concomitant diseases that could affect compliance with the protocol or interpretation of results, including significant cardiovascular disease (such as New York Heart Association Class III or IV cardiac disease, myocardial infarction within the last 6 months, unstable arrhythmias, or unstable angina) or pulmonary disease (including obstructive pulmonary disease and history of bronchospasm)
* Recent major surgery (within 4 weeks prior to the start of cycle 1), other than for diagnosis
* History or presence of an abnormal electrocardiogram (ECG) that is clinically significant in the investigator's opinion, including complete left bundle branch block, second- or third degree heart block, or evidence of prior myocardial infarction in the last 6 months
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) which requires systemic treatment. Patients may proceed with screening during treatment for infection, but systemic treatment must be completed by cycle 1 day 1.

  * If a subject has signs/symptoms suggestive of SARS-CoV-2 infection, the subject must have a negative molecular (e.g., polymerase chain reaction [PCR]) test or 2 negative antigen test results at least 24 hours apart. Subjects who do not meet SARS-CoV-2 infection eligibility criteria must be screen-failed and may only rescreen if the following have been met:

    * At least 10 days since first positive test result have passed in asymptomatic patients or at least 10 days since recovery, defined as resolution of fever without use of antipyretics and improvement in symptoms
* Positive test results for chronic hepatitis B infection (defined as positive hepatitis B surface antigen [HBsAg] serology):

  * Patients with occult or prior hepatitis B infection (defined as positive total hepatitis B core antibody and negative HBsAg) may be included if hepatitis B virus (HBV) deoxyribonucleic acid (DNA) is undetectable at the time of screening. These patients must be willing to undergo monthly DNA testing and appropriate antiviral therapy as indicated by institutional standard
* Positive test results for hepatitis C (hepatitis C virus [HCV] antibody serology testing)

  * Patients positive for HCV antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV ribonucleic acid (RNA)
* History of uncontrolled HIV

  * Patients with known diagnosis of HIV must have undetectable viral load and be on anti-retroviral therapy
* Patients with a history of progressive multifocal leukoencephalopathy
* Patients with known active central nervous system lymphoma
* Patients needing a treatment regimen which would require use of mid-cycle high dose IV methotrexate for central nervous system (CNS) prophylaxis in the opinion of the treating provider
* Pregnancy or lactation or intending to become pregnant during study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-12-07 (Actual); Primary Completion 2030-05-31 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | From the time of a subject signing consent, up until prior to Cycle 3 Day 1 (up to 42 days from Cycle 1 Day 1) or off study visit, whichever occurs earlier
  Using Common Terminology Criteria for Adverse Events version 5.0. Estimate safety and tolerability of combining epcoritamab with dose adjusted etoposide, cyclophosphamide, vincristine, doxorubicin, prednisone and rituximab.

SECONDARY OUTCOMES:
Percentage of patients that achieve a complete remission (CR) following study treatment | From the time of a subject signing consent, up until off study visit or end of treatment (Up to 18 weeks)
  A simple binary proportion will be used to estimate CR.
Progression free survival (PFS) | Up to 5 years
  Kaplan-Meier method will be used to estimate PFS.
Overall survival (OS) | Up to 5 years
  Kaplan-Meier method will be used to estimate OS.

CONTACTS AND LOCATIONS:
Overall Officials: Mengyang Di, MD, PhD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No